CLINICAL TRIAL: NCT01477099
Title: Efficacy of Toothbrushing for the Prevention of Ventilator-associated Pneumonia
Brief Title: Toothbrushing and Ventilator-associated Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Principal Investigator, Miriam Cervino, Medical Doctor, Hospital Universitario de Canarias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BRUSH-2009
Record Dates: First submitted 2011-11-16; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Toothbrushing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Toothbrushing with a manual brush (Experimental): Toothbrushing with a manual brush
  Interventions: Device: Toothbrushing with a manual brush
- No toothbrushing (No Intervention): no toothbrushing

INTERVENTIONS:
Device: Toothbrushing with a manual brush — Toothbrushing with a manual brush
  Arms: Toothbrushing with a manual brush

SUMMARY:
The hypothesis is that adding the toothbrushing to the oral care with clorhexidine 0.12% could be reduce the incidence of ventilator-associated pneumonia due to that oral cavity may be an important reservoir of pathogens that could cause pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation

Exclusion Criteria:

* edentulous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Prevention of ventilator-associated pneumonia | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Lorente, Medical, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Leonardo Lorente, San Cristóbal de La Laguna, Tenerife, Spain

REFERENCES:
- [Derived] Lorente L, Lecuona M, Jimenez A, Palmero S, Pastor E, Lafuente N, Ramos MJ, Mora ML, Sierra A. Ventilator-associated pneumonia with or without toothbrushing: a randomized controlled trial. Eur J Clin Microbiol Infect Dis. 2012 Oct;31(10):2621-9. doi: 10.1007/s10096-012-1605-y. Epub 2012 Mar 16. PMID 22422274